CLINICAL TRIAL: NCT06979336
Title: A Phase IIb, Multicenter, Double-blind, Placebo-controlled Induction Study With an Active Treatment Extension to Assess the Efficacy, Safety, and Pharmacokinetics of RO7837195 in Patients With Moderately to Severely Active Ulcerative Colitis
Brief Title: A Study to Evaluate the Efficacy, Safety, and Pharmacokinetics (PK) of RO7837195 in Participants With Moderately to Severely Active Ulcerative Colitis (UC)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GA45977; 2025-520690-39-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2025-05-15; First posted 2025-05-18 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- RO7837195 Dose Regimen 1 (Experimental): Participants will receive RO7837195 per the pre-defined dosing regimen during the 12-week induction and 40-week active treatment extension phases.
  Interventions: Drug: RO7837195
- RO7837195 Dose Regimen 2 (Experimental): Participants will receive RO7837195 per the pre-defined dosing regimen during the 12-week induction and 40-week active treatment extension phases.
  Interventions: Drug: RO7837195
- RO7837195 Dose Regimen 3 (Experimental): Participants will receive RO7837195 per the pre-defined dosing regimen during the 12-week induction and 40-week active treatment extension phases.
  Interventions: Drug: RO7837195
- RO7837195 Dose Regimen 4 (Experimental): Participants will receive RO7837195 per the pre-defined dosing regimen during the 12-week induction and 40-week active treatment extension phases.
  Interventions: Drug: RO7837195
- RO7837195 Matched Placebo/ RO7837195 (Experimental): Participants will receive RO7837195 matched placebo and RO7837195 per the pre-defined dosing regimen during the 12-week induction and 40-week active treatment extension phases, respectively.
  Interventions: Drug: RO7837195; Drug: RO7837195 Matched Placebo

INTERVENTIONS:
Drug: RO7837195 — RO7837195 will be administered as per the schedule specified in the protocol.
Drug: RO7837195 Matched Placebo — RO7837195 matched placebo will be administered as per the schedule specified in the protocol.
  Arms: RO7837195 Matched Placebo/ RO7837195

SUMMARY:
The purpose of this study is to evaluate the efficacy of RO7837195 compared with placebo in participants with moderately to severely active ulcerative colitis for whom prior treatment with conventional and/or advanced therapies has failed.

DETAILED DESCRIPTION:
This study consists of up to 5-week screening period, a 12-week induction phase, a 40-week active treatment extension, and a safety follow-up period following the last dose of study treatment. The induction phase will be placebo-controlled and after its completion, all participants will receive treatment with active study drug, regardless of the treatment response.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ulcerative colitis (UC) established at least 3 months
* Moderately to severely active UC assessed by mMS
* Inadequate response, loss of response, or intolerance to conventional or advanced therapies for UC

Exclusion Criteria:

* Prior extensive colonic resection, subtotal or total colectomy, or planned surgery for UC
* Diagnosis of Crohn's disease or indeterminate colitis
* Treatment with an advanced therapy targeted at tumor necrosis factor-like cytokine 1A (TL1a)
* Inadequate response, loss of response, or intolerance to treatment of UC with an advanced therapy targeted at IL-12 and/or IL-23

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2025-09-29 (Actual); Primary Completion 2027-08-25 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With Clinical Remission at Week 12 | At Week 12
  Clinical remission is defined as the Modified Mayo Score (mMS) of ≤ 2, including stool frequency subscore of ≤ 1, rectal bleeding subscore of 0, and endoscopy subscore of ≤ 1.

SECONDARY OUTCOMES:
Percentage of Participants With Clinical Response at Week 12 | At Week 12
  Clinical response is defined as decrease from baseline in the mMS by ≥2 and ≥ 30% reduction from baseline, with either a decrease of ≥1 in the rectal bleeding subscore or an absolute rectal bleeding subscore of ≤1.
Percentage of Participants With Endoscopic Improvement at Week 12 | At Week 12
  Endoscopic improvement is defined as a Mayo endoscopy subscore of ≤ 1.
Percentage of Participants With Endoscopic Remission at Week 12 | At Week 12
  Endoscopic remission is defined as a Mayo endoscopy subscore of 0.
Number of Participants With Adverse Events (AEs) | Up to Weeks 65
Serum Concentration of RO7837195 | Up to Weeks 65
Percentage of Participants With Anti-drug Antibodies to RO7837195 | Up to Weeks 65

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (30):
- United States (6):
  - Gastro Care Institute, Lancaster, California
  - Medical Associates Research Group, Inc., San Diego, California
  - Peak Gastroenterology Associates, Colorado Springs, Colorado
  - Clinical Research of Osceola, LLC, Kissimmee, Florida
  - Intercity Gastroenterology, Fresh Meadows, New York
  - Monroe Biomedical Research, Monroe, North Carolina
- London Digestive Disease Institute, London, Ontario, Canada
- Czechia (2):
  - PreventaMed, s.r.o., Olomouc
  - Nemocnice Slany, Slaný
- France (3):
  - CHU Saint Etienne - Hpital Nord, Saint-Étienne-de-Montluc, Pays de la Loire Region
  - CHU Clermont Ferrand - Hôpital d'Estaing, Clermont-Ferrand, Puy De Dome
  - Centre hospitalier Lyon Sud, Pierre-Bénite, Rhone
- Japan (2):
  - Fukuoka University Hospital, Fukuoka, Fukuoka
  - Takamatsu Red Cross Hospital, Takamatsu, Kagawa-ken
- Poland (14):
  - Clinsante S.C. Osrodek Badan Klinicznych, Bydgoszcz
  - Centrum Medyczne Lukamed Joanna Luka, Chojnice
  - Vita Longa Sp. z o.o., Katowice
  - MZ Badania Slowik Zymla Sp.j., Knurów
  - SOLUMED Centrum Medyczne, Poznan
  - NSZOZ Termedica Centrum Badan Klinicznych, Poznan
  - Clinical Research Center Spka z ograniczon odpowiedzialnoci Medic-R Sp.k., Poznan
  - Twoja Przychodnia-Szczecinskie Centrum Medyczne, Szczecin
  - Centrum Zdrowia MDM, Warsaw
  - Panstwowy Instytut Medyczny Ministerstwa Spraw Wewnetrznych Administracji, Warsaw
  - Provita Poliklinika sp. z o.o, Warsaw
  - Medon Clinical Research sp. z o.o, Warsaw
  - Przychodnia VISTAMED, Wroc?aw
  - ETG Zamosc, Zamość
- Chosun University Hospital, Gwangju, South Korea
- King's College Hospital, London, Greater London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing